CLINICAL TRIAL: NCT05886478
Title: Real-World Evidence Study on Brentuximab Vedotin Retreatment Outcomes of Cutaneous T-cell Lymphoma Patients
Brief Title: A Study in Adults With Cutaneous T-cell Lymphoma (CTCL) Retreated With Brentuximab Vedotin
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brentuximab-5020
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: T-Cell Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brentuximab Vedotin: Participants with CTCL who were retreated with BV after relapse will be observed retrospectively and the outcomes will be observed from June 2023 to September 2023.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The main aim of this study is to describe how effective and safe the re-treatment of adults with cutaneous T-cell lymphoma (CTCL) with brentuximab vedotin is. Another aim is to describe treatment patterns of persons with CTCL who have received brentuximab vedotin again.

No treatment will be provided during this study. Information already existing in the participants' medical charts will be reviewed and collected.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective study of participants from France, Germany, Spain and Italy with CTCL who were retreated with brentuximab vedotin (BV) after a relapse in at least two different lines of therapy. The participants will be identified from their medical charts and those who meet the eligibility criteria will be included.

The study will enroll approximately 50 participants.

This multi-center trial will be conducted in Europe. The participants are assessed after the last dose of BV for approximately 4 months and followed up for at least 12 months after the re-treatment.

ELIGIBILITY:
Inclusion criteria:

* Participant with a confirmed diagnosis of CTCL (including Mycosis fungoides (MF), Sézary syndrome (SS), Primary cutaneous CD30+ anaplastic large cell lymphoma (pcALCL) and others) who reached a complete response (CR), partial response (PR) or stable disease (SD) on a previous treatment with BV and whose disease relapsed
* Participant who was treated with BV in at least 2 lines of therapy, other treatments could have been administered in between
* Participant has received three or more cycles of BV in retreatment

Exclusion criteria:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with CTCL who were retreated with BV after relapse in France, Germany, Spain, and Italy.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) After First BV Administration | Up to approximately 12 months
ORR After Re-Treatment | Up to approximately 12 months after BV retreatment
Progression Free Survival (PFS) After First BV Administration | Up to approximately 24 months
PFS After BV Re-Treatment | Up to approximately 24 months after BV retreatment
Time to Next Treatment (TTNT) After First BV Administration (Regardless of Type of Next Treatment, i.e., BV or non-BV) | Up to approximately 16 months
TTNT After BV Re-Treatment | Up to approximately 24 months after BV retreatment
Number of Participant With Grading of Motor Neuropathy During First BV Treatment | Up to approximately 12 months
Time to Improvement of Motor Neuropathy During/ Post First BV Treatment | Up to approximately 24 months
Time to Resolution of Motor Neuropathy During/ Post First BV Treatment | Up to approximately 24 months
Number of Participants With Grading of Motor Neuropathy During BV Re-Treatment | Up to approximately 12 months after BV retreatment
Time to Improvement of Motor Neuropathy During/ Post BV Re-Treatment | Up to approximately 16 months
Time to Resolution of Motor Neuropathy During/ Post BV Re-Treatment | Up to approximately 24 months
Number of Participants With Grading of Sensory Neuropathy During First BV Treatment | Up to approximately 12 months
Time to Improvement of Sensory Neuropathy During/ Post First BV Treatment | Up to approximately 24 months
Time to Resolution of Sensory Neuropathy During/ Post First BV Treatment | Up to approximately 24 months
Number of Participants With Grading of Sensory Neuropathy During BV Re-Treatment | Up to approximately 12 months
Time to Improvement of Sensory Neuropathy During/ Post BV Re-Treatment | Up to approximately 24 months
Time to Resolution of Sensory Neuropathy During/ Post BV Re-Treatment | Up to approximately 24 months
Number of Participants With Grading of Neutropenia During First BV Treatment | Up to approximately 12 months
Number of Participants With Grading of Neutropenia During BV Re-Treatment | Up to approximately 12 months
Number of Participants With Grading of Febrile Neutropenia During First BV Treatment | Up to approximately 24 months
Number of Participants With Grading of Febrile Neutropenia During BV Re-Treatment | Up to approximately 12 months
Number of Participants With Grading of Serious Infections During First BV Treatment | Up to approximately 12 months
Number of Participants With Grading of Serious Infections During BV Re-Treatment | Up to approximately 12 months

SECONDARY OUTCOMES:
Number of Participants With Cutaneous Lymphoma Co-Medications or Strategies Used to Treat CTCL Disease | Up to approximately 12 months
Amount of BV Dose | Up to approximately 12 months
Number of Cycles of BV Administered | Up to approximately 12 months
Time Interval Between BV Administration | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- France (3):
  - Hopital Saint Andre, Bordeaux
  - Hopital Saint Louis, Paris
  - CHU Roeun, Rouen
- Germany (3):
  - Universitätsmedizin Göttingen, Göttingen
  - Klinikum Ludwigshafen, Hautklinik, Ludwigshafen
  - Universitätsklinikum Würzburg, Würzburg
- Italy (2):
  - Ospedale Maggiore Policlinico, Milan
  - AZ OSP Citta' Della Salute (Torino), Torino
- Spain (3):
  - Hospital Clinic, Barcelona, Barcelona
  - ICO Hospitalet, Barcelona, Barcelona
  - Hospital Son Espases, Palma

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/899594d64e1d4e4b?idFilter=%5B%22Brentuximab-5020%22%5D